CLINICAL TRIAL: NCT07104214
Title: Development and Validation of a Risk Prediction Model for Gastric Retention in Patients Undergoing Sedated Gastroscopy: a Multicentre Prospective Cohort Study
Brief Title: Development and Validation of a Risk Prediction Model for Gastric Retention in Patients Undergoing Sedated Gastroscopy
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Diansan Su, Chief Physician,Researcher, Zhejiang University
Other Study IDs: ZJU2025B0611
Record Dates: First submitted 2025-06-19; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Gastric Cancer Stage; Esophageal Cancer; Gastroparesis
Keywords: Gastric retention; Impaired gastric motility; Gastroparesis; Delayed gastric emptying
MeSH Terms: conditions — Esophageal Neoplasms; Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Model Development Cohort, External Validation Cohort: Model Development Cohort Definition: 3,000 patients used to identify risk factors and build the prediction mode.
  External Validation Cohort Definition: 2,000 independent patients from multiple centers to test the model's accuracy.

SUMMARY:
Gastric retention not only compromises the quality of endoscopic examination but also significantly increases the risk of reflux and aspiration in sedated patients. Aspiration of gastric contents represents a critical anesthesia-related complication during the perioperative period, carrying substantial implications for anesthetic management. With the growing volume of sedated gastroscopy procedures, predicting gastric retention has become an urgent clinical priority. This prospective study aims to establish a standardized gastric residual volume (GRV) grading system to evaluate both the volume of retained gastric contents and its contributing factors in patients undergoing upper gastrointestinal endoscopy. We will systematically assess the impact of demographic characteristics, comorbidities, and medication history on gastric emptying function. This study will facilitate establishment of an endoscopy-based simplified assessment system for gastric retention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patients scheduled for elective sedated gastroscopy or sedated gastro-colonoscopy.
* Participant provides informed consent.

Exclusion Criteria:

* Acute upper gastrointestinal bleeding (active hematemesis, melena, or confirmed UGIB within 24h).
* Emergency endoscopic procedures
* Known pregnancy or lactation
* Subjects deemed ineligible by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults scheduled for sedated gastroscopy or sedated gastro-colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed gastric emptying (defined as endoscopic gastric residual volume ≥ Grade 2) assessed by standardized endoscopic grading system | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Measurement Tool: Standardized endoscopic gastric residual volume grading system ： Grade 0：Stomach completely clean, no visible residue； Grade 1：Small amount of clear liquid (<1.5 mL/kg or <100 mL), no solid components； Grade 2：Liquid ≥1.5 mL/kg (or ≥100 mL) or small solid fragments (<5 mm)； Grade 3：Large amount of liquid (>200 mL) or significant solid residue (≥5 mm fragments) Grade 4：Visible undigested food chunks or intact food pieces Data Collection: Two physicians independently assessed gastric residue (liquid/solid), measuring volume using a graduated suction bottle, with video recordings archived for third-party review.
  Statistical Methods: The incidence (%) of gastric retention (≥Grade 2) was calculated. Multivariate logistic regression analyzed risk factors, and ROC curves evaluated the model's predictive performance (AUC).

SECONDARY OUTCOMES:
Correlation between gastric residual volume (GRV) grading and Gastroparesis Cardinal Symptom Index (GCSI) scores (range: 0-20, higher scores indicate worse symptoms) | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  The standardized Gastroparesis Cardinal Symptom Index (GCSI) was used to quantify the following core symptoms:
  Nausea (frequency & intensity): 0 (none) to 5 (severe, persistent daily).
  Vomiting (episode frequency): 0 (none) to 5 (≥3 times/day).
  Postprandial fullness (duration): 0 (none) to 5 (>4 hours).
  Early satiety (food intake limitation): 0 (normal eating) to 5 (eating <25% of usual amount).
  Statistical Analysis: The correlation between GRV grades (0-4) and the total GCSI score was assessed using Spearman's rank correlation coefficient.
Development and validation of a simplified clinical scoring system for gastric retention risk stratification (score range: 0-10, higher scores indicate higher risk) | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  Development Method: Based on multivariate logistic regression results, independent predictive factors (e.g., diabetes, GLP-1 medication use) were converted into a clinical scoring system (e.g., 1-2 points per factor).
  Validation Process:
  Discrimination: The AUC (area under the curve) of the scoring system was calculated in the validation cohort (target >0.7).
  Calibration: The Hosmer-Lemeshow test was used to assess the agreement between predicted and observed risks.
  Example Scoring Range:
  0-3 points: Low risk、4-6 points: Moderate risk、7-10 points: High risk.
Incidence of Gastric Retention in Patients Undergoing Gastroscopy | Patients will be followed for the duration of hospital stay, an expected average about 2 hours

OTHER OUTCOMES:
Incidence and risk factors of anesthesia-related adverse events in patients undergoing sedated gastroscopy | Patients will be followed for the duration of hospital stay, an expected average about 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Dr, Study Chair — Zhejiang University
Locations (3):
- China (3):
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer hospital, Hangzhou, Zhejiang
  - The Fourth Affiliated Hospital, Zhejiang University School of Medicine, Yiwu, Zhejiang

IPD SHARING:
Plan to Share IPD: No